CLINICAL TRIAL: NCT00931827
Title: Acceptability of Long-term Progestin-only Contraception in Europe
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14688; MA0801 (Other: company internal); 14239 (Other: company internal); 14177 (Other: company internal); 14176 (Other: company internal); 14016 (Other: company internal)
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Contraception
Keywords: Contraception
MeSH Terms: interventions — Levonorgestrel; etonogestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1
  Interventions: Drug: Levonorgestrel IUS (Mirena, BAY86-5028)
- Group 2
  Interventions: Drug: Implanon (Etonogestrel)

INTERVENTIONS:
Drug: Levonorgestrel IUS (Mirena, BAY86-5028) — Patients under daily life treatment receiving Mirena according to local drug information.
  Groups: Group 1
Drug: Implanon (Etonogestrel) — Patients under daily life treatment receiving Implanon according to local drug information.
  Groups: Group 2

SUMMARY:
The study examines the use of Mirena or Implanon for long-term contraception in women. The duration of therapy use is the key focus of the study. Also, any reasons for discontinuation and the safety profile will be examined. In addition, patients are asked to fill out a short questionnaire about their menstrual bleeding before and during therapy.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20-35 in good general health requesting contraception
* Women who have used short-acting hormonal contraception (combined or progestogen-only pills, vaginal ring or contraceptive patch) for at least 3 cycles immediately before entering the study and opting to change to either Mirena or Implanon for contraception
* Women who have given a written informed consent to participate in the study (if applicable)

Exclusion Criteria:

* The contraindications and warnings of the respective Summary of Product Characteristics (Mirena or Implanon) must be followed. The decision to start Mirena or Implanon has to be made clearly before the decision to include patients in the study
* Patients who are breast-feeding at time of inclusion for the study will also be excluded since breast-feeding affects the bleeding pattern

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women aged 20-35 years switching from short-acting hormonal contraception
Sampling Method: Non-Probability Sample
Enrollment: 436 (Actual)
Dates: Start 2008-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Continuation rate | At 24 months

SECONDARY OUTCOMES:
Continuation rate | At 12 months
Bleeding intensity, dysmenorrhea, and user satisfaction (questionnaires completed by patient) | Initial and after 3, 6, 12 and 24 months
Cumulative discontinuation rate for unintended pregnancy, bleeding problems, other medical reasons, for non-medical reasons | At 24 months
Incidence of Adverse Events, Serious Adverse Events | During 24 months
The return to fertility of women discontinuing the method for wish for pregnancy | 12 months after discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- Many Locations, France
- Many Locations, Ireland
- Many Locations, Slovakia
- Many Locations, United Kingdom